CLINICAL TRIAL: NCT00002190
Title: A Phase II Open-Label Exploratory Study of Saquinavir + Zidovudine + Lamivudine in HIV Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 229N; NV15114
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-07

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Saquinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Saquinavir
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To explore the antiviral efficacy, tolerability and safety of saquinavir plus zidovudine plus lamivudine.

DETAILED DESCRIPTION:
A total of 30 patients receive the triple drug regimen saquinavir plus zidovudine plus lamivudine until the completion of the analysis after at least 4 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV antibody positive.
* CD4 count >= 150 and <= 500 cells/mm3.

Exclusion Criteria

Prior Medication:

Excluded:

* Prior antiretroviral therapy.
* Prior protease inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Davies Med Ctr / c/o HIV Institute, San Francisco, California
  - Pacific Oaks Med Group / Rsch & Scientific Investigation, Sherman Oaks, California
  - Columbia Presbyterian Med Ctr, New York, New York